CLINICAL TRIAL: NCT03414606
Title: Social Behavior in Depression
Acronym: HLGDep
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Normal University (Other)
Collaborators: Huilongguan Hospital (Unknown)
Responsible Party: Principal Investigator, ma, yina, Principal Investigator, Beijing Normal University
Other Study IDs: HLGdepression
Record Dates: First submitted 2018-01-22; First posted 2018-01-30 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the project, investigators basically plan to test the difference in social behavior and social cognition between depressive patients and healthy individuals. To test this, investigators plan to use traditional or novel behavioral experiment paradigms to target various behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18 and 60
* Education experience above high school
* Score for Hamilton's Depression Scale >=17
* Diagnosis of depression through Scid

Exclusion Criteria:

* Undergoing electric shock treatment in 3 months
* Excluding those who with bipolar disorder
* Excluding those who with postpartum depression
* Excluding those who with hysteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals diagnosed with depression and healthy control
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-16 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Prosocial behavior | Baseline
  The prosocial behavior will be assessed by conventional economic games, including dictator game, message game, and ultimatum game.
Cognitive flexibility | Baseline
  Cognitive flexibility will be assessed by psychological cognitive paradigm, i.e. reversal learning paradigm. The participants will be asked to choose the item with high probability to win reward.
Valuation of social information | Baseline
  The valuation of social information was measured by psychological paradigm, developed from animal studies, called "pay-per-view". The participants will be asked make decision about more social information or more monetary reward.
Optimism bias | Baseline
  Participants will complete two sessions of life event estimation, i.e. estimating their likelihood of experiencing each event on a self-paced basis.
Emotion recognition | Baseline
  After viewing a video, participants will be asked to judge the person's attitude in the video. Through this paradigm, investigators could test emotional bias in social interaction in depressive patients.
Model-free & model-based tendency | Baseline
  Participants will be asked to complete a two-stage task, by choosing the stimuli with high probability to obtain reward.

CONTACTS AND LOCATIONS:
Overall Officials: Yina Ma, Doctor, Study Chair — Beijing Normal University
Locations (1):
- Huilongguan Hospital, Beijing, China